CLINICAL TRIAL: NCT05163704
Title: Safe Sedation of Children During Radiological Examinations
Brief Title: Dexmedetomidine Sedation in Children Before MRI Examinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Sandra Diaz Ruiz, Associate Professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MR-Dexdor
Record Dates: First submitted 2021-11-17; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Deep Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI Dexmedetomidine sedation (Other): Drug used: Dexmedetomidine. Given in increments of 0.2 ml at the time with atomizer (MAD Nasal™, Wayne Pennsylvania). Administered by radiology staff.
  Dose 1 of nasal dexmedetomidine: 4 mcg/kg max 200 mcg Dose 2 of nasal dexmedetomidine: 2 mcg/kg max 100 mcg
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is a beneficial sedative for children. It provides a sedation equivalent to a natural deep sleep with negligible respiratory effects. Administration via the nose provides better absorption and faster impact effect. The drug does not taste and does not sting when administered.
  Other Names: Intranasal spray

SUMMARY:
Dexmedetomidine, has been used in the past 4-5 years as an alternative sedation method for children at the pediatric radiology department in order to reduce the waiting lists and the use of general anesthesia with its risks and side effects in magnetic resonance and computed tomography examinations.

DETAILED DESCRIPTION:
Dexmedetomidine is a beneficial sedative for children. It provides a sedation equivalent to a natural deep sleep with negligible respiratory effects. The sedative can be administered intravenously, intranasally or buccally. Administration via the nose provides better absorption and faster impact effect. The drug does not taste and does not sting when administered. Dexmedetomidine is easy to administer and results in fewer anxious and upset patients. Monitoring the patient during the waiting period after application, during the examination itself and during the recovery period is a must. The study shows that a drug that can be administered intranasally, is practical and not invasive and means that the patient's anxiety is reduced, which can be considered an effective and safe method. Within the MRI unit at the pediatric radiology department, it has been necessary to design new routines for simple sedation, mainly due to the increased need for MRI examinations on children. Anesthesia and radiology staff have developed a new way of working where Dexmedetomidine is given nasally. These routines, including the referral flow, patient flow and staffing, have now been well established for about four years with very good results. The patient, who does not need to be fasting before the examination, receives a spray dose of the drug in the nose, falls into a deep sleep, is examined and then sleeps for about 30 minutes to an hour under supervision before returning home. It is the anesthetist who assesses which children are suitable for the type of sedation and radiology staff who are responsible for drug administration / monitoring of the patient. A preparation room is dedicated to these patients.

The patients were scheduled according to regular routine for dedicated Dexmedetomidine sedation sessions and only scans with an anticipated duration of maximum 1 hour were selected for the Dexmedetomidine protocol.

Following admission to the radiology out-patient clinic it was confirmed that the child's health condition had not changed since the last visit to the pediatrician, that there were no signs of an ongoing respiratory infection. No fasting requirements was used, and the child could eat and drink freely until arrival to the radiology clinic . Following admission and a brief period for the child to adapt to the new environment, heart rate (HR), pulse oximetry saturation and non-invasive blood pressure (NIBP) was recorded. The clinic was thereafter noticed from the MRI suite approximately 30 minutes prior to the scheduled time for the MRI examination. At this time the radiographer administered intra-nasal Dexmedetomidine. The child was then left with the accompanying caregiver/-s and the clinic nurses and checked after 15-20 min on how the sedation process evolved.

When called for, the patient was transported to the MRI suite together with the caregivers. If asleep or clearly sedated the child was placed in the MRI and prepared for the examination, which included ear plugs and noise protection earphones. A pulse oximeter probe was attached to monitor oxygenation and pulse rate. Noninvasive blood pressure or supplemental oxygen was not used during the scan since this may, according to previous clinical experience, awake the patients during the scanning procedure.

If the patient was deemed not sedated enough, an additional dose of intranasal Dexmedetomidine was administered and the child was left alone with the caregiver to allow it to settle following the administration. The child was thereafter continuously supervised by the radiographer. As the child developed a sufficient level of sedation the patient was then transferred to the scanner in the way described immediately above.

If two doses of intranasal Dexmedetomidine did not provide the desired result, the child was cancelled and rescheduled for a dedicated general anesthesia MRI session at a later occasion.

Following the scanning procedure, the ear plugs, and the noise protectors were removed, and the child was transferred from the gantry to the patient stretcher in the MRI suite area. Patients were allowed to wake up spontaneously during this process, no active efforts to wake them up were made. The pulse oximeter was left in place throughout transfer and until the child was deemed sufficiently alert in the clinic. When the child appeared reasonably awake and stable, a consensus decision made by the radiology personnel and the caregivers, the child and caregivers could return home. Before this, a new set of HR, NIBP and saturation was recorded.

ELIGIBILITY:
Inclusion Criteria:

• Healthy children, according to the American Society of Anesthesiologists (ASA) risk classification. Children with ASA risk class 1 or 2 were selected by the anesthesiologist as suitable for radiographer handled sedation with Dexmedetomidine.

Exclusion Criteria:

* Children with significant comorbidity (ASA risk class 3 or 4) that were deemed to need presence of an anesthesia team (anesthesiologist plus certified anesthesia nurse) for safety reasons.
* Children that due to the specific nature of the MRI scan would need a general anesthetic to provide a secure airway (e.g., laryngeal mask airway or endotracheal intubation) during the scan (e.g., mild neck manipulation to assess cervical instability in Mb Down patients, multiple different MRI investigations requested or need for apnea).
* Children that present minimal cold symptoms the day of imaging.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1091 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in oxygen desaturation using Dexmedetomidine to replace general anesthesia prior to magnetic resonance imaging examination | Pre-sedation, during examination and post-sedation up to 24 weeks
  During the scan the following important safety issue was followed: oxygen desaturation (SpO2 < 95 %) monitored by pulse oximetry. Low SpO2 was defined as a level below the mean value for age. If the SpO2 dropped below these levels, appropriate actions were taken (i.e., contact anesthesiologist).
  Since no fasting restrictions is part of the Dexmedetomidine-MRI protocol, specific attention was paid to the potential occurrence of regurgitation of stomach contents and/or aspiration during the entire sedation period.
  Pre- and post-sedation SpO2 (recorded in the radiology clinic pre- vs. post-scan) was compared to identify any negative effects on HR and NIBP during the early post-scan phase.
Changes in heart rate using Dexmedetomidine to replace general anesthesia prior to magnetic resonance imaging examination | Pre-sedation, during examination and post-sedation up to 24 weeks
  During the scan the following important safety issue was followed: heart rate, monitored by pulse oximetry. Low heart rate was defined as a level below the mean value for age. If the heart rate dropped below these levels, appropriate actions were taken (i.e., contact anesthesiologist).
  Pre- and post-sedation heart rate (recorded in the radiology clinic pre- vs. post-scan) were compared to identify any negative effects on SpO2 and NIBP during the early post-scan phase.
Changes in non-invasive blood preassure using Dexmedetomidine to replace general Changes in NIBP using Dexmedetomidine to replace anesthesia prior to magnetic resonance imaging examination | Pre-sedation, during examination and post-sedation up to 24 weeks
  During the scan the following important safety issue was followed: NIBP monitored. Low or high systolic and/or dyastolic blood preassure was defined according the mean value for age. If any of parameters changed below/above the normal levels for age, appropriate actions were taken (i.e., contact anesthesiologist).
  Pre- and post-sedation NIBP (recorded in the radiology clinic pre- vs. post-scan) were compared to identify any negative effects on HR and SpO2 during the early post-scan phase.

SECONDARY OUTCOMES:
Assessment of image quality using Dexmedetomidine as a sedative for children undergoing MRI examination | After sedation through study completion, an average of 1.5 years
  All scans were reviewed by a certified pediatric MRI radiologist. Scan quality was classified as optimal, slight sub-optimal but of acceptable quality to answer the diagnostic question or inadequate to allow any acceptable radiologic interpretation.

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Dillner, MD PhD, Study Chair — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
We keep working to find the lowest dose of Dexmedetomidine as possible to reach a satisfactory sedation dose. We can share our preliminary results with the actual doses but we think that lower doses can be used to obtain the same good results.
Supporting Information: Study Protocol
Time Frame: 2022
Access Criteria: Protocol with doses and way of administration will shares with radiology and anesthesiology departments who wants to implement the method. Contact could be establish by e-post and local visit for demonstration will be available. Contact with the Central contact person and the Central contact back-up could be made.

REFERENCES:
- [Result] Pansini V, Curatola A, Gatto A, Lazzareschi I, Ruggiero A, Chiaretti A. Intranasal drugs for analgesia and sedation in children admitted to pediatric emergency department: a narrative review. Ann Transl Med. 2021 Jan;9(2):189. doi: 10.21037/atm-20-5177. PMID 33569491
- [Result] Zhang Y, Zhang R, Meng HY, Wang MX, Du SZ. [Efficacy and safety of intranasal dexmedetomidine premedication for children undergoing CT or magnetic resonance imaging: a systematic review and meta-analysis]. Zhonghua Er Ke Za Zhi. 2020 Apr 2;58(4):314-318. doi: 10.3760/cma.j.cn112140-20191224-00830. Chinese. PMID 32234139
- [Result] Li L, Zhou J, Yu D, Hao X, Xie Y, Zhu T. Intranasal dexmedetomidine versus oral chloral hydrate for diagnostic procedures sedation in infants and toddlers: A systematic review and meta-analysis. Medicine (Baltimore). 2020 Feb;99(9):e19001. doi: 10.1097/MD.0000000000019001. PMID 32118711
- [Result] Mondardini MC, Amigoni A, Cortellazzi P, Di Palma A, Navarra C, Picardo SG, Puzzutiello R, Rinaldi L, Vitale F, Zito Marinosci G, Conti G. Intranasal dexmedetomidine in pediatrics: update of current knowledge. Minerva Anestesiol. 2019 Dec;85(12):1334-1345. doi: 10.23736/S0375-9393.19.13820-5. Epub 2019 Oct 14. PMID 31630510
- [Result] Uusalo P, Guillaume S, Siren S, Manner T, Vilo S, Scheinin M, Saari TI. Pharmacokinetics and Sedative Effects of Intranasal Dexmedetomidine in Ambulatory Pediatric Patients. Anesth Analg. 2020 Apr;130(4):949-957. doi: 10.1213/ANE.0000000000004264. PMID 31206433
- [Derived] Karlsson J, Lewis G, Larsson P, Lonnqvist PA, Diaz S. Intranasal dexmedetomidine sedation for paediatric MRI by radiology personnel: A retrospective observational study. Eur J Anaesthesiol. 2023 Mar 1;40(3):208-215. doi: 10.1097/EJA.0000000000001786. Epub 2022 Dec 22. PMID 36546479